CLINICAL TRIAL: NCT04486222
Title: Therapeutic Effect of Accelerated Bilateral Repeated Transcranial Magnetic Stimulation on Geriatric Depression: a Prospective Double-blind, Randomized Controlled Trial
Brief Title: Accelerated Bilateral rTMS on Geriatric Depression
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: difficulty in recruiting suitable candidate
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Taiwan University Hospital, Yun-Lin Branch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 201910101RIND
Record Dates: First submitted 2020-07-15; First posted 2020-07-24 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2021-05

CONDITIONS: Transcranial Magnetic Stimulation; Depressive Disorder, Major
Keywords: repeated transcranial magnetic stimulation; geriatric depression; anxiety; cognitive impairment; heart rate variability
MeSH Terms: conditions — Depressive Disorder, Major; Anxiety Disorders; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): The experimental group would receive an rTMS course with high-frequency stimulation (10Hz) at left DLPFC (120% motor threshold, 40 trains, 1600 pulses) followed by low-frequency (1Hz) inhibition at right DLPFC (120% motor threshold, 10 trains, 1200 pulses), two sessions daily with a 1.5-hour inter-session interval (L't active-R't active-1.5 hr-L't active-R't active), five days a week, and two weeks in total.
  Interventions: Device: Repeated Transcranial Magnetic Stimulation
- Standard Treatment Group (Active Comparator): The standard treatment group would receive an rTMS course with high-frequency stimulation (10Hz) at left DLPFC (120% motor threshold, 40 trains, 1600 pulses) followed by sham inhibition at right DLPFC (1Hz, 10 trains, 1200 pulses); after a 1.5-hour inter-session interval, a sham session would be administered at left and right DLPFC (L't active-R't sham-1.5 hr-L't sham-R't sham. The course would be applied five days a week, and two weeks in total.
  Interventions: Device: Repeated Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Repeated Transcranial Magnetic Stimulation — Magstim® Super Rapid² Transcranial Magnetic Stimulation System

SUMMARY:
This study aims to evaluate the efficacy of accelerated bilateral repetitive transcranial magnetic stimulation (rTMS) on major depression, anxiety, cognitive function and physiological parameters in elderly depressive patients.

DETAILED DESCRIPTION:
Repeated transcranial magnetic stimulation (rTMS) is a non-invasive brain stimulation treatment, showing good therapeutic effect to medicine treatment-refractory patients. Recent studies suggested bilateral DLPFC might be effective to geriatric depression. Accelerated treatment course was reported to have similar therapeutic effect and safety profile with traditional course. The investigators hypothesize accelerated bilateral rTMS is effective to geriatric depression and comorbid anxiety.

Cognitive impairment and decreased parasympathetic tone are common in patients with major depression. The investigators hypothesize cognitive function and physiological indicators improve after accelerated bilateral rTMS.

In this single-center, prospective double-blind, randomized, active-controlled trial, the investigators aim to recruit 100 patients older than 60 years, without neurocognitive disorders, and refractory to one or more antidepressants. The experimental group would receive an rTMS course with high-frequency stimulation at left DLPFC followed by low-frequency inhibition at right DLPFC, two sessions daily, five days a week, and two weeks in total. The standard treatment group would receive an rTMS course with high-frequency stimulation at left DLPFC as standard treatment parameters. Mood, cognition and physiological markers would be monitored every week. The primary outcome is response and remission rate of major depression measured by Hamilton Rating Scale for Depression.

ELIGIBILITY:
Inclusion Criteria:

* age between 60-85 years
* literate and received basic education for at least 2 years
* diagnosis of major depressive disorder, without psychotic features, according to DSM-5
* have a score of 20 or greater on the 17-item Hamilton Depression Rating Scale
* failed to achieve clinical response by at least 1 antidepressant trial of sufficient dosage for at least 4 weeks
* psychoactive agents were in stable doses before randomization

Exclusion Criteria:

* active suicide plans or attempts; or suicide attempts in the last 12 months
* diagnosis of schizophrenia or bipolar disorder according to DSM-5
* have DSM-5-confirmed substance use disorder (excluding tobacco) in the last 3 months
* have delirium, major neurocognitive disorder or MMSE < 24
* current use of bupropion >300 mg/day, tricyclic antidepressant, clozapine, chlorpromazine, foscarnet, ganciclovir, ritonavir, theophylline or anti-epileptic agents excluding benzodiazepines
* history of severe head trauma, epilepsy, multiple sclerosis, stroke, brain tumors, intracranial aneurysm, active intracranial infection, increased intracranial pressure, metallic implants in the brain, major brain surgery or major neurological diseases
* with a cardiac pacemaker or defibrillator
* received rTMS treatment before

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2020-11-23 (Actual); Primary Completion 2022-12-21 (Actual); Study Completion 2022-12-21 (Actual)

PRIMARY OUTCOMES:
Degree of Change in 17-item Hamilton Depression Rating Scale (HAM-D 17) | day 1, day 5, day 12, day 19
  HAM-D 17 is a scale rating the severity of depression, covering emotional, cognitive and somatic symptoms of depression. Higher scores indicate higher severity. Response to treatment is defined as ≥ 50% decrease in HAM-D 17; remission is defined as ≤ 7 points in HAM-D 17.

SECONDARY OUTCOMES:
Degree of Change in Hamilton Anxiety Rating Scale (HAM-A) | day 1, day 5, day 12, day 19
  HAM-A is a scale rating the severity of anxiety, covering emotional, cognitive and somatic symptoms of anxiety. Higher scores indicate higher severity.
Degree of Change in Mini-Mental State Examination (MMSE) | day 1, day 5, day 12, day 19
  MMSE is a wildly-used tool to evaluate several cognitive function domains.
Degree of Change in Stroop Test | day 1, day 5, day 12, day 19
  Task 1 (word phase) requests a subject to say a color name string (red, green, blue) printed in black; Task 2 (color phase) requests a subject to say the printed colors (red, green, blue) of letter "x" string; Task 3 (interference phase) requests a subject to say the printed colors of a string of color names (red, green, blue).
Degree of Change in Trail Making Test | day 1, day 5, day 12, day 19
  Task 1 requests a subject to connect a sequence of 25 consecutive numbers regardless of their colors; Task 2 requires a subject to connect 25 consecutive numbers in alternative colors.
Degree of Change in Verbal Fluency Test | day 1, day 5, day 12, day 19
  This test requests a subject to speak as many names of vegetables, fishes or fruit as possible in 45 seconds.
Degree of Change in Physiological Parameters | day 1, day 5, day 12, day 19
  ProComp5 Infiniti (SA7525) Biofeedback System would be used. Heart rate variability, skin conductance, body temperature and respiratory rate would be measured.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychiatry, National Taiwan University Hospital, Yun-Lin Branch, Douliu, Taiwan

IPD SHARING:
Plan to Share IPD: No